CLINICAL TRIAL: NCT00184626
Title: Safety and Efficacy of Insulin Glargine Versus Biphasic Insulin Aspart 30/70 or Biphasic Insulin Aspart 30/70 in Combination With Metformin in Subjects With Type 2 Diabetes.
Brief Title: Comparison of Insulin Glargine Versus Biphasic Insulin Aspart 30/70 or Biphasic Insulin Aspart 30/70 in Combination With Metformin in Subjects With Type 2 Diabetes.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIASP-1594
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70; Insulin Glargine; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: biphasic insulin aspart
Drug: insulin glargine
Drug: metformin

SUMMARY:
This trial is conducted in Asia. The aim of the trial is to compare the glycaemic control of Insulin glargine versus Biphasic Insulin Aspart 30/70 or Biphasic Insulin Aspart 30/70 in combination with metformin in subjects with Type 2 Diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Body mass index equal to or lesser than 35.0 kg/m2
* Currently treated with oral hypoglycaemic drug

Exclusion Criteria:

* Known hypoglycaemia unawareness or recurrent major hypoglycaemia as judged by the Investigator
* Any condition that the Investigator and/or the Sponsor feel would interfere with trial participation or evaluation of results

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2004-09-10 (Actual); Primary Completion 2005-10-24 (Actual); Study Completion 2005-10-24 (Actual)

PRIMARY OUTCOMES:
HbA1c | Measured at end of treatment (26 weeks)

SECONDARY OUTCOMES:
safety variables
other glycemic variables
Fasting plasma glucose value

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Istanbul, Turkey (Türkiye)

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com